CLINICAL TRIAL: NCT03552497
Title: The Potential of Radiomics to Differentiate Between Malignant and Benign Bosniak 3 Renal Cysts.
Acronym: BIII
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Maastricht University (Other)
Collaborators: University of California, San Francisco (Other); Stanford University (Other); Erasmus Medical Center (Other); Memorial Sloan Kettering Cancer Center (Other); University of Sao Paulo General Hospital (Other); University Hospital, Aachen (Other)
Responsible Party: Sponsor
Other Study IDs: BIIIP_18
Record Dates: First submitted 2018-05-29; First posted 2018-06-12 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Renal Cyst Complex
Keywords: Radiomics; Bosniak classification; Renal cell carcinoma; Medical imaging
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Radiomics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Radiomics — The high-throughput extraction of large amounts of quantitative image features from radiographic medical images

SUMMARY:
More than 200,000 new cases of renal cancer are diagnosed in the world each year, with more than 63,000 new cases in Europe alone. Of those, renal cell carcinoma (RCC) is the most common type in adults, making up more than 90% of the cases. Deciding on the benign or malignant nature of some RCC on the basis of medical images (CT, MRI, US) is an issue, which often leads to unnecessary surgery, morbidity and costs.

A categorization for renal cysts was introduced in the late 1980s known as the Bosniak classification. The Bosniak classification system classifies them into groups that are benign (I and II) and those that need surgical resection (III and IV), based on specific imaging features. However, defining the malignancy of category III lesions still remains a challenge. Though Bosniak classification for renal cysts is used worldwide and underwent a number of modifications, Bosniak III cysts still have almost a 1:1 chance of being malignant. So the problem is that approximately half of the Bosniak category III cystic lesions prove to be benign after surgery.

The proposed project aims to develop a quantitative image analysis (QIA) based multifactorial decision support system (mDSS) capable of classifying renal cysts with high accuracy into benign or malignant status, thus reducing the amount of unnecessary surgeries performed. Using standard-of-care CT images and clinical parameters, the customized DSS will then guide experts in planning a safe and effective diagnostic and treatment strategy for all RCC patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent contrast-enhanced CT-Scan, with radiological findings suggestive of Bosniak 3 renal cyst and have available results for pathology analysis of the cyst.

Exclusion Criteria:

* CT-Scans that are reformatted or secondary.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with renal cysts classified as bosniak 3 in one of the collaborating institutes.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-08-07 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
malignancy classifier | 1 year
  Machine learning algorithm that can differentiate between malignant and beingn bosniak 3 renal cysts.

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided